CLINICAL TRIAL: NCT05516836
Title: Addressing Post-COVID-19 Musculoskeletal Symptoms Through Telemedicine
Brief Title: Addressing Post-COVID-19 Musculoskeletal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Eleuterio Atanasio Sánchez Romero, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Addressing post-COVID-19
Record Dates: First submitted 2022-08-21; First posted 2022-08-26 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Telemedicine; Musculoskeletal Disease; SARS-CoV-2; Pain; COVID-19; Exercise
Keywords: Telemedicine; SARS-CoV-2; Rehabilitation; Therapeutic exercise
MeSH Terms: conditions — Musculoskeletal Diseases; Pain; COVID-19; Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be conducted between March 2023 and November 2024 in 62 male and female patients impacted by post-COVID-19 musculoskeletal symptoms who will undergo a multicomponent rehabilitation program, together with an intervention and a follow-up using programmed telemedicine sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercise program + Telemedicine (Experimental): The multicomponent exercise program lasted 6 weeks with sessions twice a week for a total of 12 sessions. It will have a duration of forty minutes in which the first five and the last five will be performed at a constant load of 5% of its maximum load corresponding to the "warm-up" and "return to calm". Individualized respiratory physiotherapy exercises (diaphragmatic stimulation, positive expiratory pressure exercises, alveolar retraining and strengthening of the inspiratory musculature) will also be performed.
  A once a week telemedicine session will be carried out with the case group only before the face-to-face sessions, consisting of education, respiratory exercise, mobility and stretching, giving them a place to provide feedback and re-evaluate patients mid-treatment and will be aimed at assessing improvement and improving therapeutic adherence
  Interventions: Other: Multicomponent exercise program; Other: Tele-health primary care rehabilitation program
- Multicomponent exercise program (Active Comparator): The multicomponent exercise program lasted 6 weeks with sessions twice a week for a total of 12 sessions. It will have a duration of forty minutes in which the first five and the last five will be performed at a constant load of 5% of its maximum load corresponding to the "warm-up" and "return to calm". Individualized respiratory physiotherapy exercises (diaphragmatic stimulation, positive expiratory pressure exercises, alveolar retraining and strengthening of the inspiratory musculature) will also be performed.
  Interventions: Other: Multicomponent exercise program

INTERVENTIONS:
Other: Multicomponent exercise program — Each exercise session will have a duration of forty minutes in which the thirty minutes of intervallic work will be distributed as follows: twenty seconds until reaching 60% of their maximum load in the first seven sessions, adding five watts each day until reaching 80% of their maximum load in the fourteen sessions and seventy seconds of rest at 20% of their maximum load.
  At the end of the sessions, strengthening exercises will be performed with elastic bands, adapting their resistance according to the characteristics of the patients, of the lower limbs and of the upper limbs. Individualized respiratory physiotherapy exercises (diaphragmatic stimulation, positive expiratory pressure exercises, alveolar retraining and strengthening of the inspiratory musculature) will also be performed.
Other: Tele-health primary care rehabilitation program — A once a week telemedicine session will be carried out with the case group only before the face-to-face sessions, consisting of education, respiratory exercise, mobility and stretching, giving them a place to provide feedback and re-evaluate patients mid-treatment and will be aimed at assessing improvement and improving therapeutic adherence.
  Arms: Multicomponent exercise program + Telemedicine

SUMMARY:
The purpose of the study will be to evaluate the effect of a rehabilitation program on the improvement of patients with post-COVID-19 musculoskeletal symptoms, as well as to quantify the impact of telemedicine that evaluates the evolution of pain, functionality, and quality of life.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted in 100 patients with post-COVID-19 musculoskeletal symptoms who will undergo a multicomponent rehabilitation program, together with an intervention and a follow-up using programmed telemedicine sessions. Data will be collected on the improvement of functional capacity and quality of life, in addition to assessing the evolution of musculoskeletal symptomatology, as well as pain and psychological variables. The telemedicine sessions will improve user adherence and follow-up, and the results are expected to be disseminated to the scientific community during and after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Need to be post-COVID-19 patients (ICU or non-ICU)
* Musculoskeletal symptoms
* Be of adult age (over 18 years)

Exclusion Criteria:

* Myocardial infarction
* Uncontrolled arrhythmia
* Recent pulmonary thromboembolism
* Terminal illness
* Patients undergoing lower limb unloading
* Lower or upper limb fractures in the last three months
* Severe pain (score greater than 7 on the VAS of 10 points)
* Suffering from the previous pathology that causes neuromuscular weakness
* Be younger than 18 and older than 65 years old
* Influenced by medication that does not allow assessment of the real muscular functionality of the patient
* Patients with cognitive impairment that would prevent them from understanding and collaborating in the performance of the rehabilitation program plus telemedicine
* Patients with cardiorespiratory instability and uncontrolled arterial hypertension
* Systemic illness (tumor and rheumatologic diseases)
* Recent unrelated trauma
* Limiting psychiatric pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Manual grip strength | Change from base line and at the end of each of the six weeks
  Grip strength will be measured in the affected hand and in the healthy hand (measuring the maximum grip strength). For this measurement, Handgrip strength averaging the result of three attempts with the dominant hand using a Baseline© model pear dynamometer
Quality of life according to Short- Form 36 Questionnaire (SF - 36) | Change from base line and at the end of each of the six weeks
  SF - 36 is an instrument to asses health - related quality of life, this evaluates eight spheres (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health) scored from zero to 100, where 100 is equivalent to no disability and zero is equivalent to maximum disability.
Assessment of exercise capacity | Change from base line and at the end of each of the six weeks
  Exercise capacity will be measured with a six-minute walking test (6MWT), a sub-maximal exercise test which consists of the patient walking for six minutes along a 30 - meter corridor with two cones marking the distance to be covered while being given a series of cues.
COPD Assessment Test (CAT) | Change from base line and at the end of each of the six weeks
  CAT is an eight item questionnaire to assess: cough, sputum, chest tightness, breathlessness, activity limitation, confidence leaving home, sleep and energy scored from zero to 4 in each item, zero corresponds to the least affected and 5 to the most affected

SECONDARY OUTCOMES:
Dyspnea using the modified Medical Research Council dyspnea scale (mMRC) | Change from base line and at the end of each of the six weeks
  This scale assess dyspnea in activities of daily living scored from 0 (absence of dyspnea during intense exercise) to 4 (dyspnea prevents the patient from leaving the house or appears with tasks such as dressing or undressing)
Assessment of perceived pain | Change from base line and at the end of each of the six weeks
  The numerical pain intensity scale adds a numerical graduation where 1 is no pain and 10 is the worst pain imaginable. The confidence and reliability of this scale has been approved and validated in different studies.
STAI (State-Trait Anxiety) | Change from base line and at the end of each of the six weeks
  Questionnaire composed of 20 items with 4 points each that evaluate "state anxiety" (transitory emotional condition influenced by environmental factors that decrease or increase anxiety) and another 20 that evaluate "trait anxiety" (personality factor that predisposes to suffer or not suffer anxiety). The 2-part score ranks patients at a percentile to the general population. The higher the score, the greater the anxiety. It is one of the most widely used tools in research to measure levels of general anxiety.
TSK (Tampa Scale for Kinesiophobia) | Change from base line and at the end of each of the six weeks
  7 items, 4 points each where higher scores indicate higher levels of fear of movement.
Beck II (Depression) | Change from base line and at the end of each of the six weeks
  A 21-item scale used to assess the severity of depression. The patient has to select for each item the response alternative that best reflects his/her state during the last week. The total score is obtained by adding up the values of the selected items, which range from 0 to 3. The commonly accepted cut-off points for grading intensity/severity are as follows: 0 to 9, no depression; 10 to 18, mild depression; 19 to 29, moderate depression, and ≥ 30 points, severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Hugo Villafañe, PhD, Study Chair — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Eleuterio A. Sánchez Romero, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez-Romero EA, Garcia-Barredo-Restegui T, Martinez-Rolando L, Villafane JH, Galan-Fraguas A, Jurado-Molina R, Cuenca-Zaldivar JN, Soto-Goni XA, Martinez-Lozano P. Addressing post-COVID-19 musculoskeletal symptoms through pulmonary rehabilitation with an evidence-based eHealth education tool: Preliminary results from a pilot randomized controlled clinical trial. Medicine (Baltimore). 2025 Mar 7;104(10):e41583. doi: 10.1097/MD.0000000000041583. PMID 40068080